CLINICAL TRIAL: NCT06479551
Title: Comparative Effects of High and Moderate Intensity Resistance Training on Strength, Power and Muscle Soreness in Young Football Players
Brief Title: Comparative Effects of High and Moderate Intensity Resistance Training in Young Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0490 maria
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Sports Physical Therapy
Keywords: Footballer; Muscle soreness; Power; Resistance Training; Sprint
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: A (Experimental): 13 participants will be in experimental group giving them High intensity-low volume resistance training protocol of 4 reps and 2 sets comprising 90% of 1 RM parallel back squats for six weeks measure all values before giving them protocol and after protocol.
  Interventions: Other: high intensity-low volume resistance training
- Control Group: B (Experimental): 13 participants will be in control group giving them moderate intensity-high volume resistance training training protocol of 8 reps and 3 sets comprising 80% of 1 RM parallel back squats for six weeks measure all values before giving them protocol and after protocol.
  Interventions: Other: Moderate intensity-high volume resistance training

INTERVENTIONS:
Other: high intensity-low volume resistance training — 13 participants will be in experimental group giving them High intensity-low volume resistance training protocol of 4 reps and 2 sets comprising 90% of 1 RM parallel back squats for six weeks measure all values before giving them protocol and after protocol.
  Arms: Experimental Group: A
Other: Moderate intensity-high volume resistance training — 13 participants will be in control group giving them Moderate intensity-high volume resistance training of 8 reps and 3 sets comprising 80% of 1 RM parallel back squats for six weeks measure all values before giving them protocol and after protocol.
  Arms: Control Group: B

SUMMARY:
Football playing is an intermittent sport requiring high intensity dynamic movements, such as acceleration, sprinting and jumping. Higher levels of strength and power are crucial for young football players. Overuse includes using a muscle too much, too soon before warming up, or too often in gym, Tension or stress can cause muscle soreness. DOMS is thought to be due to temporary muscle damage and inflammation for which the most common trigger appears to be eccentric exercises. Exercise induced muscle damage DOMS is considered a type1 muscle strain injury that has a pain free period of one day. Muscle soreness peaks between one to two days. The objective of this study is to compare the effects of high intensity-low volume (HRT) versus moderate intensity-high volume resistance training (MRT) on strength, power and muscle soreness in young football players.

Study will be a randomized clinical trial, conduct at Pakistan football federation Lahore through convenient sampling techniques. Sample size will be calculated by using G-power. Randomization will be done by Lottery method. Participants will be divided into two groups. Group A will receive High intensity resistance training and Group B will receive moderate intensity resistance training Strength will be calculated by 1RM and sprint test . Power will be measured by vertical and horizontal jump. Muscle soreness and fatigue will be measured by Hooper and MacKinnon questionnaire. Data will be analyzed by SPSS version 25

DETAILED DESCRIPTION:
The objective of my study is to compare the effects of high and moderate intensity resistance training on strength, power and muscle soreness in young football players

ELIGIBILITY:
Inclusion Criteria:

* Male and female players

  * Age 18-24yrs
  * Player with minimum 1-year experience of football
  * Muscle soreness value shouldn't be below normal.
  * Value on Hooper and Mackinnon Questionnaire should be from 1-3.
  * A minimum score of 3-4 in lower extremity functional scale
  * Fatigue shouldn't regress the normal.(45)

Exclusion Criteria:

* History of lower limb musculoskeletal injuries in last 3months

  * Fracture since last 6months
  * Taking drugs or ergogenic supplement
  * Neurological systems are not intact(dermatomes and myotomes)
  * A minimum score of in lower extremity functional scale.(65, 66)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Hooper and Mackinnon Questionnaire | six weeks
  This questionnaire was used to measure muscle soreness and fatigue .It comprised of five Questions covering fatigue, sleep,level of muscle soreness and psychological well-being. were measured before and after the intervention session ,with reliability of 0.86 with minimum measurement error it had a strong construct validity.(67)
Vertical and Horizontal Jump | six weeks
  It is a common test used to gauge athletic performance as well as an exercise for increasing strength and endurance. Athletes compete in the track and field long jump, which tests their strength, speed, and agility as they try to jump as far as they can from a takeoff point. Horizontal jump has reliability of 0.90(0.00) and vertical jump has reliability of 0.86(0.00) will be exhibiting refined concurrent validity.(68)
1RM, Sprint Test | six weeks
  Its reliability was of (ICC 0.90:CV 4.0%) measurement error 5.1 kg and ICC 0.96, measurement error 3.2 kg, respectively) was resulting with good construct validity. hese assessments are frequently used to evaluate an athlete's performance and monitor their development over time in athletic and fitness contexts.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan football federation Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Currier BS, Mcleod JC, Banfield L, Beyene J, Welton NJ, D'Souza AC, Keogh JAJ, Lin L, Coletta G, Yang A, Colenso-Semple L, Lau KJ, Verboom A, Phillips SM. Resistance training prescription for muscle strength and hypertrophy in healthy adults: a systematic review and Bayesian network meta-analysis. Br J Sports Med. 2023 Sep;57(18):1211-1220. doi: 10.1136/bjsports-2023-106807. Epub 2023 Jul 6. PMID 37414459
- [Background] Askew GN. Adaptations for extremely high muscular power output: why do muscles that operate at intermediate cycle frequencies generate the highest powers? J Muscle Res Cell Motil. 2023 Jun;44(2):107-114. doi: 10.1007/s10974-022-09640-2. Epub 2023 Jan 11. PMID 36627504
- [Background] Edouard P, Nunes JP, Koral J, Thornton JS, Kemp JL, Gronwald T. Just start and keep training! What is the best resistance training prescription for strength and hypertrophy? Br J Sports Med. 2023 Sep;57(18):1161-1162. doi: 10.1136/bjsports-2023-107234. Epub 2023 Jul 5. No abstract available. PMID 37407091
- [Background] Shah A, Bordoni B. Anatomy, Bony Pelvis and Lower Limb, Gluteus Medius Muscle. 2023 Feb 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557509/ PMID 32491441
- [Background] Khan IA, Bordoni B, Varacallo MA. Anatomy, Bony Pelvis and Lower Limb: Thigh Gracilis Muscle. 2023 Apr 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538229/ PMID 30855817
- [Background] Granger CJ, Cohen-Levy WB. Anatomy, Bony Pelvis and Lower Limb: Posterior Tibial Nerve. 2023 May 23. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK546623/ PMID 31536230
- [Background] Thomakos P, Spyrou K, Katsikas C, Geladas ND, Bogdanis GC. Effects of Concurrent High-Intensity and Strength Training on Muscle Power and Aerobic Performance in Young Soccer Players during the Pre-Season. Sports (Basel). 2023 Mar 6;11(3):59. doi: 10.3390/sports11030059. PMID 36976945
- [Background] Champ CE, Carpenter DJ, Diaz AK, Rosenberg J, Ackerson BG, Hyde PN. Resistance Training for Patients with Cancer: A Conceptual Framework for Maximizing Strength, Power, Functional Mobility, and Body Composition to Optimize Health and Outcomes. Sports Med. 2023 Jan;53(1):75-89. doi: 10.1007/s40279-022-01759-z. Epub 2022 Sep 29. PMID 36175646